CLINICAL TRIAL: NCT00539799
Title: Corticosteroids in the Maintenance Therapy of Proliferative Lupus Nephritis: a Randomized Pilot Study
Brief Title: Steroids in the Maintenance of Remission of Proliferative Lupus Nephritis
Acronym: SIMPL
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Local pharmacy unwilling to comply with study protocol
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A091040; EUDRACT: 2007-003923-20
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Lupus Nephritis
Keywords: systemic lupus erythematosus; lupus nephritis
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Long-term low-dose prednisolone (5 - 7.5 mg/day)
  Interventions: Drug: prednisolone
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: prednisolone — 5 - 7.5 mg/day
  Arms: 1
Drug: Placebo — Matched placebo to prednisolone
  Arms: 2

SUMMARY:
There is debate as to whether long-term low-dose steroids such as prednisolone help to suppress relapses of systemic lupus erythematosus (SLE) in patients who are in remission from their lupus nephritis. If low-dose prednisolone reduces relapses, these beneficial effects may be counter-balanced by the long-term side-effects associated with prednisolone. This pilot study will determine the feasibility of conducting a larger randomized control trial that will answer the question of whether or not long-term low-dose prednisolone (5 - 7.5 mg/day) reduces the flares of SLE in patients with previous lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18 years
* diagnosis of SLE by ACR criteria
* diagnosis of proliferative lupus nephritis (ISN/RPS class III or IV)
* currently on prednisolone (5 to 20 mg/day)
* in partial or complete remission for at least 3 months

Exclusion Criteria:

* currently pregnant
* in end-stage renal failure
* receiving corticosteroids for an indication other than lupus nephritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)

PRIMARY OUTCOMES:
Feasibility (recruitment rate and protocol adherence) | 12 months

SECONDARY OUTCOMES:
1) time to major renal and non-renal relapses of SLE 2) time to minor relapses of SLE 3) health related quality of life 4) adverse events/side-effects 5) accrual of SLE related organ damage 6) renal function | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: David Jayne, MD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust; Michael Walsh, MD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom